CLINICAL TRIAL: NCT06438770
Title: Predicting Independent Gait After Stroke: External Validation of a Multivariable Prediction Model
Brief Title: Prediction of Gait After Stroke; an External Validation
Status: Completed | Type: Observational
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Principal Investigator, Martina Betschart, PhD, Physiotherapist, Clinical Specialist, Kantonsspital Winterthur KSW
Other Study IDs: 2020-01966
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: prediction model; external validation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational study is to perform a temporal and geographical external validation of the EPOS (Early Prediction of Outcome after Stroke) model for the prediction of independent gait after stroke. The EPOS model measures the early presence of leg strength on the affected side and sitting ability to predict recovery of independent walking six months after stroke. Compared to the EPOS model development study, the prediction time point of independent gait in this study will be three months rather than six months post-stroke and the patients will be more heterogeneous. Due to the differences in the new cohort, it is expected that the performance of the models will be lower than in the development cohort, but still be adequate.

DETAILED DESCRIPTION:
Worldwide, stroke is the second leading cause of death and is also the third leading cause of death and disability combined. According to the Global Burden of Disease, Injuries, and Risk Factors Study (GBD) by the Collaborator Network on the topic of stroke, the absolute number of incidence strokes and their deaths have steadily increased in recent years. The most important risk factors include high blood pressure, a high body-mass index, high plasma glucose, fine dust pollution and smoking. In Switzerland, an average of 20'423 people suffered a stroke per year between 2016 and 2020. Due to the growth and ageing of the population, the number of hospitalizations due to cardiovascular diseases is increasing, but deaths have decreased over time. According to a recent study, 75% of stroke survivors are able to walk independently after three months. On average, independent walking is achieved six days post-stroke whereby stroke severity is most strongly associated with recovery of gait.

In recent years, a large number of studies have been published showing that prognosis is of growing interest in stroke rehabilitation. Medical prognostic models are used to inform patients and their families about the course of their disease and to plan possible treatments. Early prognosis of recovery after stroke enables early discharge planning and efficient use of health care resources. In addition, therapy goals can be realistically formulated and thus recommendations for care or adaptations of the home environment can be made. Currently, prognostic models are rarely used in clinical practice. This is partly because most of the models have not been externally validated, which is a prerequisite for implementation in practice. External validation involves using new data from a similar population to investigate the generalizability of the model. In summary, a good and useful prognostic model should be accurate, generalizable and ideally clinically effective.

A narrative review described six prognostic models for independent gait after stroke. Only three of these models measure predictor and outcome variables at a specifically defined time point: the Australian model, the TWIST model and the EPOS model. The Australian model and the TWIST model have been updated but not externally validated and the EPOS model has been externally validated once. According to the review above, the EPOS model seems to be a promising model for predicting independent gait after a stroke. This is due to the early and fixed time point of simple and fast clinical tests as well as the prognosis time point of six months. The EPOS model shows that early presence of lower limb strength and sitting ability can predict recovery of independent walking six months after stroke. Predictive variables were measured using the Trunk Control Test with the item "sitting balance" (TCT-s) and the Motricity Index leg score (MI leg). The dependent outcome variable was the Functional Ambulation Categories (FAC). In the external validation, the dependent outcome variable FAC was measured after three months. The results show good performance of the model from the third day onwards for predicting independent gait three months after stroke.

In summary, these findings raise the question of whether the use of the EPOS model in post-stroke patients within the first 72 hours is accurate and generalizable for predicting independent walking three months after stroke. Although this first external validation shows promising results, further external validation studies need to be undertaken before the model can be applied in clinical practice. The aim of this study is to perform a temporal and geographical external validation of the EPOS prediction model for independent gait after stroke. Compared to the development study, this study will be conducted in Switzerland and the prediction of independent gait will be based on the time point of three months rather than six months post-stroke. In addition, all post-stroke patients will be included, regardless of the type of stroke, the affected circulation or positive stroke history. Furthermore, patients with pre-existing comorbidities are also being considered, as long as they were ambulatory before the stroke.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or older
2. having suffered an ischemic or hemorrhagic stroke, confirmed by computerized tomography and/ or magnetic resonance imaging
3. being unable to walk independently (FAC < 4) within 72 hours
4. giving written informed consent to participate

Exclusion Criteria:

1. not able to walk independently before hospital admission (FAC < 4)
2. clinically significant comorbidities that prevent walking ability
3. deficits in cognition or communication, so consent cannot be given for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: admitted to hospital with an acute stroke
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Functional Ambulation Categories (0-5 points, higher scores being better) | 3 months poststroke
  functional gait

OTHER OUTCOMES:
Trunk Control Test (0-100 points, higher scores being better) | within 72 hours poststroke
  trunk movement and control
Motricity Index - lower extremity subscale (0-100 points, higher scores being better) | within 72 hours poststroke
  lower extremity limb strength

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland

REFERENCES:
- [Background] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721
- [Background] Kennedy C, Bernhardt J, Churilov L, Collier JM, Ellery F, Rethnam V, Carvalho LB, Donnan GA, Hayward KS. Factors associated with time to independent walking recovery post-stroke. J Neurol Neurosurg Psychiatry. 2021 Jul;92(7):702-708. doi: 10.1136/jnnp-2020-325125. Epub 2021 Mar 17. PMID 33737383
- [Background] Ramspek CL, Jager KJ, Dekker FW, Zoccali C, van Diepen M. External validation of prognostic models: what, why, how, when and where? Clin Kidney J. 2020 Nov 24;14(1):49-58. doi: 10.1093/ckj/sfaa188. eCollection 2021 Jan. PMID 33564405
- [Background] Moons KG, Royston P, Vergouwe Y, Grobbee DE, Altman DG. Prognosis and prognostic research: what, why, and how? BMJ. 2009 Feb 23;338:b375. doi: 10.1136/bmj.b375. No abstract available. PMID 19237405
- [Background] Kwah LK, Herbert RD. Prediction of Walking and Arm Recovery after Stroke: A Critical Review. Brain Sci. 2016 Nov 2;6(4):53. doi: 10.3390/brainsci6040053. PMID 27827835
- [Background] Altman DG, Vergouwe Y, Royston P, Moons KG. Prognosis and prognostic research: validating a prognostic model. BMJ. 2009 May 28;338:b605. doi: 10.1136/bmj.b605. No abstract available. PMID 19477892
- [Background] Langerak AJ, McCambridge AB, Stubbs PW, Fabricius J, Rogers K, Quel de Oliveira C, Nielsen JF, Verhagen AP. Externally validated model predicting gait independence after stroke showed fair performance and improved after updating. J Clin Epidemiol. 2021 Sep;137:73-82. doi: 10.1016/j.jclinepi.2021.03.022. Epub 2021 Mar 31. PMID 33812010
- [Background] Kwah LK, Harvey LA, Diong J, Herbert RD. Models containing age and NIHSS predict recovery of ambulation and upper limb function six months after stroke: an observational study. J Physiother. 2013 Sep;59(3):189-97. doi: 10.1016/S1836-9553(13)70183-8. PMID 23896334
- [Background] Veerbeek JM, Van Wegen EE, Harmeling-Van der Wel BC, Kwakkel G; EPOS Investigators. Is accurate prediction of gait in nonambulatory stroke patients possible within 72 hours poststroke? The EPOS study. Neurorehabil Neural Repair. 2011 Mar-Apr;25(3):268-74. doi: 10.1177/1545968310384271. Epub 2010 Dec 26. PMID 21186329
- [Background] Stinear CM, Smith MC, Byblow WD. Prediction Tools for Stroke Rehabilitation. Stroke. 2019 Nov;50(11):3314-3322. doi: 10.1161/STROKEAHA.119.025696. Epub 2019 Oct 15. No abstract available. PMID 31610763
- [Background] Smith MC, Barber AP, Scrivener BJ, Stinear CM. The TWIST Tool Predicts When Patients Will Recover Independent Walking After Stroke: An Observational Study. Neurorehabil Neural Repair. 2022 Jul;36(7):461-471. doi: 10.1177/15459683221085287. Epub 2022 May 18. PMID 35586876
- [Background] Veerbeek JM, Pohl J, Held JPO, Luft AR. External Validation of the Early Prediction of Functional Outcome After Stroke Prediction Model for Independent Gait at 3 Months After Stroke. Front Neurol. 2022 May 2;13:797791. doi: 10.3389/fneur.2022.797791. eCollection 2022. PMID 35585839
- [Background] Smith MC, Barber PA, Stinear CM. The TWIST Algorithm Predicts Time to Walking Independently After Stroke. Neurorehabil Neural Repair. 2017 Oct-Nov;31(10-11):955-964. doi: 10.1177/1545968317736820. Epub 2017 Nov 1. PMID 29090654
- See also: Schweizerisches Gesundheitsobservatorium — https://ind.obsan.admin.ch/
- See also: Bundesamt für Statistik — https://www.bfs.admin.ch/bfs/de/home/statistiken/gesundheit/gesundheitszustand/krankheiten/herz-kreislauf-erkrankungen.html